## The 9-Box Performance Management Framework: Impacts on Body Weight Regulation and Exercise Behaviors in Graduate Students

## Informed consent form for weight loss health management of graduate students

## Dear participants:

Hello! We are inviting you to join a management trial called the "Graduate Student Weight Loss Challenge". This study aims to explore effective weight loss methods tailored for graduate students and their impact on improving physical health. The 9-week program requires participants to complete tasks according to the weight loss protocol designed by our research team throughout the intervention period.

## Rights and obligations of participants

Voluntary Participation: You have the right to voluntarily decide whether to participate in this trial. Your decision will not affect any of your rights and interests at school; Withdrawal at Any Time: You may choose to withdraw at any stage of the study without giving reasons. Privacy Protection: Your personal information will be strictly confidential, and test data will be processed anonymously without disclosing your identity.

Your Rights: Your research record will contain a unique code used exclusively by the project team for identification purposes. All data storage devices are password-protected, accessible only to authorized members of the project management team. The results of this study may be published in academic publications, journals, or news reports. Your name and other personally identifiable information will not be used for these purposes. Participation in the informed consent form is voluntary. If you decline to participate for any reason, you are not obligated to sign it.

If you have any questions, confusion or complaints about your participation in this study, or have any questions about your rights, you may contact the contact person below this consent form.

Contact: Chen Lei Tel: 17886719603

Informed consent: I have been informed of the purpose, process and possible risks of this trial. All my questions have been answered satisfactorily. I understand that my participation is voluntary and that I can withdraw at any time without adverse effects. The following signature indicates my voluntary consent to participate in this management.

| Signature of | participant: | Date: | vear | month | day |
|---------------|--------------|----------|---------|-------|-----|
| Digitature or | participant. | <br>Date | _ y car | | uay |